CLINICAL TRIAL: NCT04368611
Title: Emergency Laparoscopic Cholecystectomy With Low Pressure Pneumo-peritoneum in Cardiopulmonary Risk Patients: Fundus First Cholecystectomy VS Calot First Cholecystectomy .Randomized Controlled Trials.
Brief Title: Emergency Laparoscopic Cholecystectomy With Low Pressure Pneumo-peritoneum in Cardiopulmonary Risk Patients: Fundus First Cholecystectomy VS Calot First Cholecystectomy .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: lap cholecystectomy 1
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Laparoscopy; Biliary Disease
Keywords: laparoscopy; cholecystectomy
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fundus first cholecystectomy (Active Comparator): start with fundus dissection then complete the dissection
  Interventions: Procedure: start with fundus
- Calot first dissection (Active Comparator): start and complete the dissection by dissection of Calot triangle
  Interventions: Procedure: calot first dissection

INTERVENTIONS:
Procedure: start with fundus — fundus first dissection then complete cholecystectomy as usual
  Arms: fundus first cholecystectomy
Procedure: calot first dissection — start dissection by calot approach
  Arms: Calot first dissection

SUMMARY:
Introduction:

Laparoscopic cholecystectomy is the usual approach in dealing with cholithiasis that greatly replace open approach even in acute emergency gall bladder diseases. Laparoscopic approach has great advantages than open approach but the biliary injuries are higher in laparoscopic approach than open approach. Laparoscopic approach is condemned for many years in cardiopulmonary risk patients because of its adverse impacts on cardiopulmonary systems. Performing laparoscopic cholecystectomy with low pressure pneumoperitoneum may be effective in treatment of acute gall bladder disease but with fundus first approach than classical Calot first approach.

Aim: compare between initial Fundus first cholecystectomy followed by Calot dissection VS Calot only cholecystectomy in Emergency laparoscopic cholecystectomy with low pressure pneumo-peritoneum in cardiopulmonary risk patients as regard intraoperative data and postoperative complications.

Patients and methods:

This study prospective randomized controlled study was conducted on 470 cases with acute cholecystitis, biliary colic, mucocele and pyocele of gall bladder in emergency general surgery department. Patients were divided into 2 groups, Group A: fundus first group (235cases) and Group B (235cases): classical Calot first approach.

DETAILED DESCRIPTION:
1. INTRODUCTION Introduction of laparoscopy in management of cholithiasis gave a great push to dealing with this disease. The advancement of laparoscopic cholecystectomy had greatly evolved in the last years making laparoscopic cholecystectomy is the commonest operation performed within field of gastrointestinal tract surgery and almost replaced open cholecystectomy.[1] [2]

   After introduction of laparoscopic cholecystectomy, many advantages the patients gained over open cholecystectomy as small operative wounds with minimal postoperative pain and infection and hence rapid discharge from hospital. Other advantages are better cosmosis, earlier resumption of oral feeding and rapid restoration of daily activity and work. [3]

   Although laparoscopic cholecystectomy had many advantages over open approach yet, many disadvantages emerged after the wide spread use of laparoscopic cholecystectomy as higher incidence of bile duct injuries that may reach 0.3-0.8% that may increase in acute emergent cases. This is a grave problem that may cause mortality to the patients. [4]Strasberg gave us the best solution up till now and the way to avoid injury to biliary tract. [5].Other complications the patients may face after laparoscopic cholecystectomy are organ injury; vascular injury and obstructive jaundice from missed stone in common bile duct during the operation. [6]

   About 30% of patients undergo laparoscopic cholecystectomy are elderly patients with cardiopulmonary risks [7]

   Co2 insufflation into the peritoneal cavity exerts bad effects on cardiac and respiratory systems and may worsen the condition of cardio-pulmonary risk patients. Pneumo-peritoneum with CO2 causes splintage of the diaphragm, hypercarbia with arrhythmias, compression of main abdominal vasculature (Inferior Vena Cava and abdominal aorta) and stretch of the peritoneal cavity with consequent parasympathetic irritation causing baradycardia.[8][9][10][11][12].

   Head up position during laparoscopic cholecystectomy exerts good effect on lung but bad effects on heart as it decreases venous return and hence cardiac output. Also, the head up position increases adrenaline level in the blood that lead to vasoconstriction of blood vessels that increase peripheral resistance and decrease cardiac output and increases load on myocardium.[13][14] [15]

   No randomized studies have compared fundus first laparoscopic cholecystectomy with low pressure pneumoperitoneum with Calot first dissection cholecystectomy in cardiopulmonary risk patients with urgent laparoscopic cholecystectomy.

   The aim of this study was to evaluate and compare the outcome of urgent LC using either fundus first approach or Calot classic approach in cardiopulmonary risk patients as regard morbidity and mortality.
2. THE AIM OF THE WORK The aim of this study was to evaluate and compare the outcome of urgent laparoscopic cholecystectomy under low pressure Pneumo-peritoneum using either fundus first approach and Calot classic approach in cardiopulmonary risk patients as regard morbidity and mortality.
3. Patients and methods Study design: Prospective Randomized controlled clinical study. Study place: our study was conducted in the surgical emergency unit of our University Hospitals.

Study period: March 2015 to March 2018. Source of data: Patients admitted with clinical diagnosis of acute cholecystitis, biliary colic, mucocele or pyocele of gall bladder in patients with cardiopulmonary diseases.

Sample size: A total of 470 patients with a clinical diagnosis of acute cholecystitis, biliary colic, mucocele or pyocele of gall bladder in patients with cardiopulmonary diseases.

Sampling method: simple random sample with a balance Method of sample size calculation: Sample size calculated to be 235 at each group based on operation time difference between conventional and funds first group from previous paper with 80% power of study and 95% confidence interval. Ref Cengiz, Y., Lund, M., Jänes, A. et al. Fundus first as the standard technique for laparoscopic cholecystectomy. Sci Rep 9, 18736 (2019). https://doi.org/10.1038/s41598-019-55401-6

Patient selection criteria:

A. Inclusion criteria:

1. Age: any age.
2. Sex: Male and Non pregnant female.
3. Patients with cardiopulmonary diseases.
4. Patients who diagnose acute cholecystitis not improving on medical treatment for 48 hours.
5. Patients with biliary colic, mucocele of gall bladder and pyocele of gall bladder.
6. American Society of Anesthesiologist's (ASA) score: grade I, II, III.

Exclusion criteria:

1. ASA grade IV
2. Patients refuse surgery.
3. Documented Liver disease.
4. Previous percutaneous cholecystostomy
5. Cases not tolerated CO2 insufflation from the start.

Preoperative work up: All patients included in the study underwent:

1. Full clinical examination: pain in right hypochondrium radiated to right shoulder, local examination revealed tenderness in right hypochondrium or mass and fever.
2. Ultrasonography: thick edematous wall of gall bladder distended gall bladder or stone impacted in gall bladder neck.
3. Blood investigations :leukocytosis
4. Liver Function Tests.
5. Chest x-ray
6. ECG and cardiac Echocardiography.

Patients are divided into 2 groups:

Group A (n = 235): patients underwent laparoscopic cholecystectomy with low pressure pneumoperitoneum and initial fundus first cholecystectomy followed by dissection of Calot triangle.

Group B (n=235): patients underwent laparoscopic cholecystectomy with low pressure pneumoperitoneum and Calot first cholecystectomy from the start.

Efforts to decrease bias in the study:

1. For pretrial bias: Good Define objectives. Risk and outcome .Select patients on probability sample with adequate sample size. Define confound factors and avoid it
2. To avoid during trial bias: Standardize reaction and management of patients blindly-Objective data use rather than subjective-Good handling of data- plan designed for drop out
3. To avoid after trial bias: Suitable statistical analysis used-Good and carefully interpretation-Control of confound

Methods:

The patients were given general anesthesia. Nasogastric and urinary bladder catheters were inserted to ensure the stomach and bladder were empty. Through the periumbilical incision, A Hasson technique was used and a trocar is introduced to the abdomen under vision. Pneumoperitoneum was created 8-10 mm Hg. The camera was introduced and the abdominal cavity inspected. A 10 mm trocar was placed at the level of epigastrium 5 cm below xiphoid process. A third 5 mm trocar was placed just below the right subcostal margin. 4th trocar is inserted at the level of umbilicus at anterior axillary line.

Fundus first approach initial approach: we start dissection of the peritoneum at the side of gall bladder and perform dissection in inverted U shaped incision in the peritoneum covering the side and fundus of gall bladder then the gall bladder is dissected free from gall bladder bed .then the fundus of gall bladder is retracted towards easily to the right shoulder and start exposure and dissection of the Calot triangle .in this way, dissection of Calot triangle became very easy. Sometimes aspiration of the gall bladder contents helped us to grasp the fundus.

Calot triangle first dissection: we started dissection at gall bladder neck. Adhesions to omentum, colon, duodenum or stomach are pulled away by blunt and diathermy dissection. Dissection continued very close to gall bladder wall. Identification of Calot triangle helped us to recognize the anatomy. Cystic duct and cystic artery are dissected free and clipped and divided. Then the gall bladder is dissected free from the liver. The gallbladder bed was inspected for hemostasis which was achieved by coagulation. The gallbladder was removed from the abdomen through the epigastric port. Irrigation and suction of the bed was performed and a drain is put in gall bladder bed. Under vision, all ports were removed. The umbilical incision was closed in layers with Vicryl No 1 and subcuticular with prolene three zero.

Outcome measures:

Primary outcomes

1. Mortality (90-day mortality and mortality at maximal follow-up).
2. Postoperative complications: early (hemorrhage, bile leak, wound infection) and late complications (biliary stricture)

4. Port site hernia Secondary outcomes

1. Conversion to open cholecystectomy.
2. Total hospital stay.
3. Intra-operative findings (duration of operation, intra-operative bleeding and iatrogenic injuries)
4. Return to work.

ELIGIBILITY:
Inclusion Criteria:

* Age: any age.
* Sex: Male and Non pregnant female.
* Patients with cardiopulmonary diseases.
* Patients who diagnose acute cholecystitis not improving on medical treatment for 48 hours.
* Patients with biliary colic, mucocele of gall bladder and pyocele of gall bladder.
* American Society of Anesthesiologist's (ASA) score: grade I, II, III.

Exclusion Criteria:

* ASA grade IV
* Patients refuse surgery.
* Documented Liver disease.
* Previous percutaneous cholecystostomy
* Cases not tolerated CO2 insufflation from the start.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
duration of operation in minutes | 2 hours
  time taken to complete the surgery in minutes

SECONDARY OUTCOMES:
stricture of the biliary tract | 2 years
  stenosed bile duct that induce jaundice on laboratory investigations

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Alsaied Alnaimy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No